CLINICAL TRIAL: NCT02916654
Title: Sucrosomial Iron Supplementation in Anaemic Patients With Celiac Disease Not Tolerating Oral Ferrous Sulfate
Brief Title: Sucrosomial Iron in Patients With Celiac Disease and IDA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33_2014
Record Dates: First submitted 2016-09-21; First posted 2016-09-27 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Celiac Disease; Iron Deficiency Anemia
MeSH Terms: conditions — Celiac Disease; Anemia, Iron-Deficiency | interventions — sucrosomial iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sulphate iron (Active Comparator): patients administered with sulphate iron
  Interventions: Drug: Sulphate iron
- sucrosomial iron (Experimental): patients administered with sucrosomial iron
  Interventions: Dietary Supplement: sucrosomial iron

INTERVENTIONS:
Dietary Supplement: sucrosomial iron — administration of sucrosomial iron
  Arms: sucrosomial iron
Drug: Sulphate iron — administration of sulphate iron
  Arms: sulphate iron

SUMMARY:
Sucrosomial iron (Sideral® Forte) is a preparation of ferric pyrophosphate conveyed within a phospholipid membrane associated with ascorbic acid, is a new-generation oral iron which shows a high gastrointestinal absorption and high bioavailability with a low incidence of side effects due to lack of any direct contact with intestinal mucosa. In comparison with the other standard oral iron preparations, sucrosomial iron seems to be a promising new strategy of iron replacement in CD patients.

ELIGIBILITY:
Inclusion Criteria:

* proven celiac disease
* iron deficiency anemia

Exclusion Criteria:

* other autoimmne diseases
* pregnancy psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda, Milan, MI, Italy